CLINICAL TRIAL: NCT07380464
Title: A New Classification System for Lymph Nodes in Colon Cancer: The Prognostic Significance of the Anatomical Distribution of Metastatic Lymph Nodes and the Number of Tumor Deposits
Status: Completed | Type: Observational
Sponsor: Cai Zerong (Other)
Responsible Party: Sponsor-Investigator, Cai Zerong, Deputy Director of the Department, Sixth Affiliated Hospital, Sun Yat-sen University
Organization: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Other Study IDs: 2025ZSLYEC-785
Record Dates: First submitted 2026-01-22; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Colon Cancer; Tumor Deposits; Lymph Node Metastases; TNM Staging
Keywords: Colon Cancer; Lymph Node Metastases; N stage
MeSH Terms: conditions — Colonic Neoplasms; Extranodal Extension; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- No metastasis
- Non-skip metastasis without tumor deposits
- No metastasis or non-skip metastasis with tumor deposits，Skip metastasis without tumor deposits
- Skip metastasis with tumor deposits, All-station metastasis regardless of tumor deposits

SUMMARY:
This study aims to investigate the prognostic significance of LNM distribution and establish a new classification system integrating both nodal quantity and anatomical location.The main question it aims to answer is:

Does the new N staging based on lymph node metastasis patterns and cancer nodules provide a more accurate prediction of the prognosis of colon cancer patients compared to the AJCC N staging? The relevant clinical characteristics, treatment processes, postoperative pathological data and post-discharge prognosis information of the enrolled patients were collected through the follow-up offices and the medical record system. The data were analyzed. The main research endpoints were: overall survival (the time between the initial surgery and death or the last follow-up); disease-free survival (the time between the initial surgery and disease metastasis, recurrence or death).

ELIGIBILITY:
Inclusion Criteria:

* Definite diagnosis of primary colon adenocarcinoma via auxiliary examination or pathology.
* No distant metastasis (M0) confirmed by preoperative imaging or intraoperative findings.
* No prior neoadjuvant therapy (including chemotherapy, radiotherapy, immunotherapy, or targeted therapy).
* Underwent initial radical resection for colon cancer.
* Available data on lymph node counts for all three stations.

Exclusion Criteria:

* Intraoperative or postoperative pathology confirming non-malignant tumors (including carcinoma in Tis).
* Multiple primary cancers or concurrent malignancies in other sites.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study enrolled a total of 1,500 participants between January 2010 and December 2022. Inclusion criteria were defined as follows: (1) a confirmed diagnosis of primary colon adenocarcinoma via auxiliary examination or pathology; (2) absence of distant metastasis (M0) verified by preoperative imaging or intraoperative findings; (3) initial radical colectomy; and (4) complete documentation of lymph node counts across three stations. Patients were excluded if they had received any form of neoadjuvant therapy (including chemotherapy, radiotherapy, immunotherapy, or targeted therapy) prior to surgery. Additionally, cases were excluded if intraoperative or postoperative pathology revealed non-malignant tumors (including carcinoma in Tis) or if patients presented with multiple primary cancers or concurrent malignancies in other sites.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2010-03-05 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
DFS | From the date of the initial surgery to death or disease recurrence or metastasis,assessed up to 120 months
  Disease Free Survival
OS | From the date of the initial surgery to death, assessed up to 120 months
  Overall Survival

CONTACTS AND LOCATIONS:
Overall Officials: Zerong Cai, MD, Study Director — Sixth Affiliated Hospital, Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: No
Please contact us by Email.